CLINICAL TRIAL: NCT00002115
Title: A Phase I/II Study of the Safety, Tolerance, and Pharmacokinetics of 9-(2-Phosphonylmethoxyethyl)Adenine ( PMEA; Adefovir ) in Patients With Advanced HIV Disease.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 217A; GS-92-202
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1995-11

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; Antiviral Agents; Adenine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — adefovir

INTERVENTIONS:
Drug: Adefovir

SUMMARY:
To study the safety, tolerance, pharmacokinetics, and anti-HIV effects of PMEA ( adefovir ) when administered daily by intravenous (IV) and/or subcutaneous (SC) injection in patients with advanced HIV disease.

DETAILED DESCRIPTION:
Patients receive a single IV or SC dose of PMEA daily for 4 weeks. A maximum tolerated dose will be defined for these regimens.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Other antiretroviral therapy IF on a stable dose for at least 4 weeks prior to study entry.
* Prophylactic therapy with aerosolized pentamidine, oral trimethoprim/sulfamethoxazole (Bactrim, Septra) or dapsone, and fluconazole or ketoconazole IF on a stable prophylactic regimen for at least 4 weeks prior to study entry.

Patients must have:

* HIV seropositivity.
* Elevated p24 antigen (> 40 pg/ml).
* Mean CD4 count <= 100 cells/mm3.
* Life expectancy of at least 3 months.

Prior Medication:

Allowed:

* Other prior antiretroviral therapy.
* Prophylactic therapy with aerosolized pentamidine, oral trimethoprim/sulfamethoxazole (Bactrim, Septra) or dapsone, and fluconazole or ketoconazole.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Inadequate venous access.
* Active serious infection (other than HIV infection) requiring parenteral antibiotic therapy.
* Clinically significant cardiac disease, including symptoms of ischemia, congestive heart failure, or arrhythmia.
* Psychiatric disturbance or illness that may affect compliance.
* Malignancy other than Kaposi's sarcoma.

Concurrent Medication:

Excluded:

* Investigational agents other than stavudine (d4T).
* Interferon-alpha.
* Ganciclovir.
* Foscarnet.
* Diuretics.
* Amphotericin B.
* Aminoglycoside antibiotics.
* Other nephrotoxic agents.
* Acyclovir at doses >= 2 g/day.

Prior Medication:

Excluded within 2 weeks prior to study entry:

* Investigational agents other than stavudine (d4T).
* Interferon-alpha.
* Ganciclovir.
* Foscarnet.
* Diuretics.
* Amphotericin B.
* Aminoglycoside antibiotics.
* Other nephrotoxic agents.

Excluded within 4 weeks prior to study entry:

* Systemic therapy for Kaposi's sarcoma. Substance abuse.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20

CONTACTS AND LOCATIONS:
Locations (1):
- Univ of Washington, Seattle, Washington, United States